CLINICAL TRIAL: NCT04266964
Title: Muscle Excitability Scale for Assessment of Spastic Reflexes in Spinal Cord Injury. Part II: Validity and Reliability Study
Brief Title: Validity and Reliability Study of the Muscle Excitability Scale in Spinal Cord Injury Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Jiri Kriz, MD, PhD, Clinical Professor, University Hospital, Motol
Other Study IDs: SCI_MES_2019
Record Dates: First submitted 2020-02-05; First posted 2020-02-12 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Spasticity, Muscle; Spinal Cord Injuries
Keywords: Spasticity; Spinal cord injury; Validity; Reliability
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Manual examination — With the patient in a supine position, squeeze the skinfold between your thumb and pointfinger on the inner aspect of the middle third of the thigh and on the inner aspect of the middle third of the calf.
  Place your hand under the proximal calf and the heel and move the leg into maximum flexion at the hip and knee joints. After the response, if any, is completed, move the limb back into full extension. Each of these movements lasts for one second.

SUMMARY:
The aim of the study is to verify validity and reliability of the Muscle excitability scale (MES), which has been developed to access muscle susceptibility to spasms and/or clones as part of spastic motor behavior in spinal cord injured patients.

DETAILED DESCRIPTION:
The muscle excitability scale (MES) is intended for patients after spinal cord injury. The objective is to evaluate a motor response (muscle spasms or clones) to a sensory or motor stimulus. A sensory stimulus is created by thumb and pointfinger compression of cutaneous tissue on the inside part of the middle thigh and calf. A motor stimulus is created by passive movement of the lower limb to flexion and extension. The MES grades from 0 to 4 reflect the muscle spastic or clonic tendency and the extent of this motor response (from isolated to generalized). Two investigators will examine a spastic motor behavior in 50 chronic SCI subjects using MES, Modificated Ashworth Scale (MAS) and Penn Spasms Frequency Scale (PSFS) to verify the validity and reliability of the MES.

ELIGIBILITY:
Inclusion Criteria:

* Spasticity in Spinal Cord Injury

Exclusion Criteria:

* Parallel brain injury
* Cognitive deficit affecting cooperation
* Acute infection or other sudden complication
* Recent change of antispastic medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spasticity in spinal cord injury
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Muscle Excitability Scale | through study completion, an average of 1 year
  Scoring from 0 to 4; 0 = no motor response (muscle spasm or clonus) to a tactile stimulus or passive movement; 4 = generalized motor response to both a tactile stimulus and passive movement
Modified Ashworth Scale | through study completion, an average of 1 year
  Scoring from 0 to 4; 0 = no increase in muscle tone; 4 = affected part(s) rigid in flexion or extension
Penn Spasm Frequency Scale | through study completion, an average of 1 year
  Scoring 0 to 4; 0 = no spasms; 4 = spasms occurring more than 10 times per hour

SECONDARY OUTCOMES:
Calculation of validity and reliability index of Muscle Excitability Scale | through study completion, an average of 1 year
  To determine validity, inter-rater and intra-rater reliability of the Muscle Excitability Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Kriz, MD, PhD, Principal Investigator — Spinal Cord Unit, University Hospital, Motol
Locations (2):
- Czechia (2):
  - Department of Rehabilitation and Sports Medicine, University Hospital Motol, Prague
  - Paraple Center - rehab center for SCI people, Prague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kriz J, Hlinkova Z. Muscle excitability scale - a novel tool for evaluation of spastic motor behaviors in spinal cord injury patients. In: Proceedings from the 55th ISCoS Annual Scientific Meeting; September 14-16, 2016; Vienna, Austria. Abstract 186.